CLINICAL TRIAL: NCT05431907
Title: Phase 1/2 Study Evaluating Safety and Potential Efficacy of Allocetra-OTS Via Pressurized Intra-Peritoneal Aerosol Chemotherapy as Add-on to Standard of Care Chemotherapy for Treatment of Peritoneal Metastasis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Enlivex Therapeutics RDO Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ENX-CL-04-001
Record Dates: First submitted 2022-06-08; First posted 2022-06-24 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Peritoneal Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohorts 1-2 (Experimental): Escalating doses of Allocetra-OTS up to 10 x 10^9 cells.
  Interventions: Drug: Allocetra-OTS
- Cohorts 3-4 (Experimental): Allocetra-OTS at the maximal tolerated dose.
  Interventions: Drug: Allocetra-OTS

INTERVENTIONS:
Drug: Allocetra-OTS — Allocetra-OTS is a cell-based therapy consisting of non-HLA matched allogeneic peripheral blood mononuclear cells, derived from a healthy human donor following a leukapheresis procedure, induced to an apoptotic stable state.

SUMMARY:
This is an open-label study to evaluate safety and potential efficacy of Allocetra-OTS in the treatment of patients with peritoneal metastasis as an add-on to the standard of care (SoC) chemotherapy.

DETAILED DESCRIPTION:
Pressurized Intra-Peritoneal Aerosol Chemotherapy (PIPAC) is utilized in patients with malignant dissemination to the peritoneal cavity, for the treatment of peritoneal metastasis that have a high tumor burden or are unresectable, and are unresponsive to systemic therapy.

Allocetra-OTS is an immunomodulatory cell-based therapy consisting of allogeneic peripheral blood mononuclear cells that have been modified to be engulfed by macrophages and reprogram them into their homeostatic state.

The study will evaluate the safety and potential efficacy of Allocetra-OTS in the treatment of peritoneal metastasis as an add-on to the standard of care (SoC) chemotherapy. Patients will be treated with escalating doses of Allocetra-OTS as an add-on to the chemotherapy administered via PIPAC, and in addition to systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Diagnosis of peritoneal metastasis due to any primary tumor by histopathology or cytology
* Possession of unresectable tumors (not eligible for Cytoreductive Surgery / Hyperthermic Intra-Peritoneal Chemoperfusion CRS/HIPEC).
* Adequate performance status and surgical risk
* Adequate hematopoietic, hepatic and renal function

Exclusion Criteria:

* Extraperitoneal disease.
* Bowel obstruction
* History of Liver cirrhosis with CHILD PUGH classification of B or C or signs of portal hypertension, portal vein thrombosis.
* Patient with known New York Heart Association (NYHA) class 3 or 4 symptomatic congestive heart failure, severe myocardial insufficiency, recent myocardial infarction, severe arrhythmias.
* Previous history of organ allograft or stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Number and severity of Allocetra-OTS related adverse events (AEs) and serious adverse events (SAEs) | 16 weeks
  Number and severity of Allocetra-OTS related adverse events (AEs) and serious adverse events (SAEs) during 16-week period starting from the first administration of study treatment.

SECONDARY OUTCOMES:
Best Overall Response Rates (BORR) | 16 weeks
  Best Overall Response Rates (BORR) will be comprised of clinical, radiological and pathology assessments.
Change in specific cancer markers | 16 weeks
  Change in the specific cancer markers (CEA, CA-19-9, CA-125) from baseline to each post-PIPAC assessment.
Progression-free survival (PFS) | 6 months
  Progression-free survival (PFS) assessed based on imaging data (PET/CT)
Overall Survival (OS) | 12 months
  OS up to 12 months from the first administration of study treatment.
Change in quality of life | 16 weeks
  Change in quality of life according to EORTC QLQ-CR29 from screening to 16 weeks.

OTHER OUTCOMES:
Additional Safety Endpoint: Number and severity of related AEs and SAEs throughout 6 months from the first administration of study treatment. | 6 months
  Number and severity of related AEs and SAEs throughout 6 months from the first administration of study treatment.
Exploratory Endpoint: Change in macrophages and immune cells characteristics in peritoneal fluid | 12 weeks
  Change in macrophages and immune cells characteristics in peritoneal fluid and tissues from baseline up to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Avi Nissan, MD, Principal Investigator — Department of Surgical Oncology, Sheba Medical Center
Locations (1):
- The Chaim Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No